CLINICAL TRIAL: NCT05996107
Title: A Phase 1B Study of Ribociclib Administered Concurrently With Postoperative Radiation Therapy in Patients With High-Risk, HR+/HER2- Breast Cancer
Brief Title: Study of Ribociclib Administered Concurrently With Postoperative Radiation Therapy in Patients With High-Risk, HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2022.071; HUM00231659 (Other: University of Michigan)
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: HR+/HER2-; Node positive; High-Risk breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RT + Ribociclib (Experimental): All patients will be treated with Ribociclib and standard of care radiation therapy
  Interventions: Drug: Ribociclib; Radiation: Postoperative Radiation Therapy

INTERVENTIONS:
Drug: Ribociclib — 400 mg daily with a possibly dose reduction to 200 mg daily if required
  Other Names: Kisqali
Radiation: Postoperative Radiation Therapy — 50 Gy in 25 fractions or 42.56 Gy in 16 fraction +/- 10 Gy boost including comprehensive nodal

SUMMARY:
The purpose of this research study is to determine the safety, tolerability and dose of Ribociclib when combined with adjuvant radiation in women with high-risk ER+ breast cancer.

Once enrolled on study, patients will begin treatment with Ribociclib 400 mg daily at the same time as they initiate standard of care adjuvant radiation therapy- 50 Gy in 25 fractions or 42.56 Gy in 16 fractions +/- 10 Gy boost including comprehensive nodal. Paitents will continue treatment with Ribociclib for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ER and/or PR-positive (≥ 1% positivity as determined by local pathology laboratory), HER2-negative breast cancer with > 3 lymph nodes involved on sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) OR have between 1-3 lymph nodes involved AND have T3 disease OR have between 1-3 lymph nodes involved and grade 3 breast cancer.
* Age ≥ 18
* Patients must have undergone gross total excision of all locoregional disease with negative margins (i.e. no tumor on ink). At least 21 days must elapse between surgical treatment for breast cancer and initiation of study treatment.
* Patients must have completed chemotherapy (either in neoadjuvant or adjuvant setting). If received adjuvant chemotherapy, chemotherapy must have completed at least 21 days prior to initiation of study treatment.
* Participants must have recovered (grade ≤1) from the acute effects of chemotherapy and surgical side effects following definitive breast surgery except for neuropathy and alopecia
* Adequate baseline hematologic, hepatic and renal function as indicated below:

  * Patient has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by central laboratory for eligibility):
  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug)
  * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m2 according to the Modification of Diet in Renal Disease (MDRD) formula
  * Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.
  * Aspartate transaminase (AST) < 2.5 × ULN, except for patients with liver metastasis, who are only included if the AST is < 5 × ULN
  * Alanine transaminase (ALT) < 2.5 × ULN, except for patients with liver metastasis, who are only included if the ALT is < 5 × ULN
  * Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements before the first dose of study medication:
  * Potassium
  * Magnesium
  * Total Calcium (corrected for serum albumin)
* QTcF interval at screening EKG ≤ 450ms (QT interval using Fridericia's correction).
* Mean resting heart rate 50-90 bpm (determined from the EKG).
* Ability to swallow study drug (Ribociclib).
* ECOG Performance Status 0-1 (Karnofsky > 60%).
* Availability of archival tumor tissue from surgical specimen.
* Ability to understand and willingness to sign informed consent.
* Women of childbearing potential must have confirmed negative pregnancy test (urine or serum) within 14 days of initiation of study treatment.

Exclusion Criteria:

* Prior history of radiation therapy to the chest wall and/or regional nodes is not allowed (but prior radiation therapy to other sites is permissible).
* Prior history of CDK4/6 inhibitor therapy.
* Patients who are pregnant or breastfeeding.

  • Because radiation is known to be teratogenic, women of childbearing potential must have a documented negative pregnancy test performed prior to the start of study therapy (as above) and agree to use adequate contraception (hormonal or double barrier method of birth control; vasectomized partner; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patient with distant metastases of breast cancer beyond regional lymph nodes and/or evidence of breast cancer recurrence prior to study enrollment.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  * History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft within 6 months prior to trial entry.
  * Documented cardiomyopathy.
  * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) (testing not mandatory)
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
  * Risk factors for Torsades de Pointes (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
  * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause TdP that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting trial treatment).
  * Inability to determine the QTcF interval.
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third degree AV block).
  * Uncontrolled arterial hypertension with systolic blood pressure > 160 mmHg.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, liver cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infections, active infection requiring systemic antibacterial therapy, etc.) or limit life expectancy to ≤5 years. Questions regarding inclusion of individual subjects should be directed to Drs. Cobain and Speers (ecobain@med.umich.edu and cspeers@med.umich.edu).
* Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 2 years before randomization. Note: Patients with adequately treated, basal or squamous cell skin carcinoma or curatively resected cervical cancer in situ are eligible.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the oral trial treatments (e.g. uncontrolled ulcerative diseases, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, or small bowel resection).
* Patients must not receive any additional anti-cancer therapy or investigational agents during study therapy. Anti-cancer therapies include chemotherapy and endocrine therapy.
* Patient is currently receiving any of the following substances within 7 days before randomization:

  * Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pummellos, starfruit, Seville oranges) and their juices that are known as strong inhibitors or inducers of CYP3A4/5.
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of ribociclib administered concurrently with adjuvant RT 1 month post last RT dose | up through 30 days after the last dose of study drug or radiotherapy
  Safety evaluations will be based on the incidence, intensity, and type of adverse events, and clinically significant changes in the patient's physical examination, vital signs, and clinical laboratory results. Safety variables will be tabulated and presented for all patients in the study. Exposure to study drug and reasons for discontinuation of study treatment will be tabulated.

SECONDARY OUTCOMES:
Cumulative incidence of local failure (i.e. local recurrence events) | up through 2 years after completion of protocol therapy
  Calculation of follow-up time for all endpoints for patients will begin from the date of diagnosis until documentation of local or regional recurrence for local control, any failure (local, regional, or distant) or death for recurrence-free survival, and death for overall survival.
Local failure-free survival | up through 2 years after completion of protocol therapy
  The time from diagnosis date to the first of local or regional recurrence or death. Patients who are alive and free of local regional recurrence at lat follow up will be cencored at that date.
Recurrence-free survival | up through 2 years after completion of protocol therapy
  Date of diagnosis until documentation of death. Time-dependent and will be summarized using the Kaplan-Meier method or cumulative incidence method when competing events.
Overall survival | up through 2 years after completion of protocol therapy
  Overall survival as determined by the date of diagnosis until documentation of death. Time-dependent and will be summarized using the Kaplan-Meier method or cumulative incidence method when competing events.
Disease free survival | up through 2 years after completion of protocol therapy
  Defined as the time to the first of local, regional, or distant recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Erin Cobain, MD, Principal Investigator — University of Michigan Rogel Cancer Center; Corey Speers, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health West, Wyoming, Michigan
  - UHCMC Seidman Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No